CLINICAL TRIAL: NCT05945706
Title: Evaluation of Renal Resistance Index by Doppler Ultrasonography in Patients Undergoing Arthroscopic Shoulder Surgery with Controlled Hypotension
Brief Title: Evaluation of Renal Resistive Index in Patients with Controlled Hypotension
Status: Completed | Type: Observational
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Özkan Sipahioğlu, MD, Specialist, Principal Investigator, Ankara Diskapi Training and Research Hospital
Other Study IDs: Renal Rezistif Index
Record Dates: First submitted 2023-07-05; First posted 2023-07-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Acute Kidney Injury; Hypotension, Controlled; Renal Failure; Ultrasonography, Doppler
Keywords: acute kidney injury; blood flow velocity; Renal Doppler ultrasound; Renal Resistive Index; Controlled hypotension
MeSH Terms: conditions — Acute Kidney Injury; Hypotension; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In recent studies, it has been reported that the renal resistive index is effective in detecting postoperative acute kidney injury in the early period. This study aims to evaluate the preoperative and postoperative renal resistive index variation with intraoperative controlled hypotension and research the renal resistive index's utility in the early detection of renal dysfunction that may develop after surgery.

DETAILED DESCRIPTION:
Controlled hypotension could be defined as a reduction of the systolic blood pressure to 80-90 mmHg, a reduction of mean arterial pressure (MAP) to 50-65 mmHg, or a 30% reduction of baseline MAP (1). It is frequently applied in orthopedics, neurosurgery, and ear-nose-throat surgeries to reduce blood loss and provide a good field of view to the surgeon. However, the combination of hypotension with hypovolemia may result in postoperative acute kidney injury (AKI), especially in the elderly and in patients with hypoperfusion-sensitive disease. The situation may worsen with nephrotoxic drugs.

In patients with AKI, the length of hospital stay is prolonged, and the risk of morbidity and mortality increases, so early detection of AKI is significant. Perioperative AKI diagnosis is difficult and often delayed. Although there are various tests (cystatin-c, urea, serum creatinine, creatinine clearance, etc.), there is still no early, accurate, easy-to-use AKI marker in clinical practice.

The most commonly used guidelines for AKI classification are 2004-RIFLE (Risk, Injury, Failure, Loss of kidney function, End stage renal disease), 2007-AKIN (Acute Kidney Injury Network), and 2012-KDIGO (Kidney Disease Improving Global Outcomes). Based on the validity of the RIFLE and AKIN criteria, the KDIGO guideline was developed to diagnose AKI with a straightforward definition for clinical practice.

Doppler ultrasonography is widely used in the evaluation of chronic kidney diseases. Renal resistive index (RRI), one of the Doopler-derived indices, is calculated by imaging the intrarenal (arcuate or interlobar) artery and measuring the highest systolic and lowest end-diastolic blood flow velocity using a colored Doppler. It is generally accepted that the normal value of the RRI is 0.60 ± 0.01 (mean±SD), and there is a general opinion that the upper limit of the RRI is 0.7 (2). The renal resistive index has been used for years to diagnose and follow up on various kidney diseases (evaluation of chronic renal allograft rejection, detection and management of renal artery stenosis, and chronic differential diagnosis) (3). Recent studies have reported that RRI effectively detects postoperative AKI in the early period before the criteria for AKIN are formed (4-5).

This study aims to evaluate the preoperative and postoperative renal resistive index variation with intraoperative controlled hypotension and research the renal resistive index's utility in the early detection of renal dysfunction that may develop after surgery.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* will undergo elective arthroscopic shoulder surgery
* ASA (American Society of Anesthesiologist Classification) I-II or III

Exclusion Criteria:

* Cardiac arrhythmia
* Asymmetric kidney disease
* Poor echogenicity (for imaging)
* Chronic renal dysfunction (GFR<30)
* Renal artery stenosis
* Endocarditis
* Postoperative agitation or confusion
* Postoperative polypnea >35/min or respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ASA I-II-III patients who are scheduled to undergo elective arthroscopic shoulder surgery older than 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Renal resistive index | baseline, pre-surgery
  Renal resistive index measurement by Doppler ultrasonography before anesthesia induction
Renal resistive index | immediately after the surgery under anesthesia
  Renal resistive index measurement by Doppler ultrasonography at the end of surgery under anesthesia
Renal resistive index | within 30 minutes after surgery
  Renal resistive index measurement by Doppler ultrasonography in the postanesthetic care unit

SECONDARY OUTCOMES:
serum creatinine | preoperative (baseline)
  blood serum creatinine level at admission to the hospital
serum creatinine | postoperative day 1
  blood serum creatinine level on postoperative day one
serum creatinine | postoperative day 2
  blood serum creatinine level on postoperative day two
postoperative urine output | every 6 hours for 48 hours
  postoperative urine output measurement

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ozkan Sipahioglu, MD, Principal Investigator — Ankara Diskapi Training and Research Hospital
Locations (1):
- Dıskapı Training and Research Hospital, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu N, Chen L, Liu L, Rong W. Dexmedetomidine versus remifentanil for controlled hypotension under general anesthesia: A systematic review and meta-analysis. PLoS One. 2023 Jan 17;18(1):e0278846. doi: 10.1371/journal.pone.0278846. eCollection 2023. PMID 36649357
- [Background] Tublin ME, Bude RO, Platt JF. Review. The resistive index in renal Doppler sonography: where do we stand? AJR Am J Roentgenol. 2003 Apr;180(4):885-92. doi: 10.2214/ajr.180.4.1800885. No abstract available. PMID 12646425
- [Background] Marty P, Ferre F, Labaste F, Jacques L, Luzi A, Conil JM, Silva S, Minville V. The Doppler renal resistive index for early detection of acute kidney injury after hip fracture. Anaesth Crit Care Pain Med. 2016 Dec;35(6):377-382. doi: 10.1016/j.accpm.2015.12.013. Epub 2016 Apr 28. PMID 27133237
- [Background] Bossard G, Bourgoin P, Corbeau JJ, Huntzinger J, Beydon L. Early detection of postoperative acute kidney injury by Doppler renal resistive index in cardiac surgery with cardiopulmonary bypass. Br J Anaesth. 2011 Dec;107(6):891-8. doi: 10.1093/bja/aer289. Epub 2011 Sep 22. PMID 21940396
- [Background] Viazzi F, Leoncini G, Derchi LE, Pontremoli R. Ultrasound Doppler renal resistive index: a useful tool for the management of the hypertensive patient. J Hypertens. 2014 Jan;32(1):149-53. doi: 10.1097/HJH.0b013e328365b29c. PMID 24172238